CLINICAL TRIAL: NCT02154230
Title: Effect of Sulphate-bicarbonate-calcium Water Consumption on the Body Weight and Gut Microbiota Composition in Overweight and Obese Patients Under Low-calorie Diet
Brief Title: Sulphate-bicarbonate-calcium Water, Body Weight and Gut Microbiota
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: failure to enroll
Sponsor: University of Roma La Sapienza (Other)
Collaborators: TERME DI CHIANCIANO Spa, Italy (Unknown)
Responsible Party: Principal Investigator, STEFANO GINANNI CORRADINI, MD, PhD, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2488/14.06.2012
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Overweight; Obesity
Keywords: weight loss; sulphate-bicarbonate-calcium water; gut microbiota; body composition; bile salts
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- sulphate-bicarbonate-calcium water and low-calorie diet (SW-D) (Experimental): Experimental arm: Those patients assigned to this interventional arm of the study will be asked to follow a low-calorie diet. For the first 12 weeks, the diet will cover only basal metabolism expenditure ± 10%. At the end of this 12 weeks, for the following 12 weeks, patients will follow a maintenance diet which will cover both basal metabolism and physical activity expenditure. Patients will be invited to maintain the same level of physical activity preceding enrollment throughout the entire study period. During the first 4 weeks these patients will be asked to drink every morning, before breakfast, within 30 minutes, 500 mL of "Acqua Santa di Chianciano"® at room temperature.
  Interventions: Dietary Supplement: "Acqua Santa di Chianciano"® (sulphate-bicarbonate-calcium water)
- tap water and low-calorie diet (TW-D) (Active Comparator): Active comparator: Those patients assigned to this interventional arm of the study will be asked to follow the same low-calorie diet of the experimental arm. During the first 4 weeks these patients will be asked to drink every morning, before breakfast, within 30 minutes, 500 mL of Rome tap water at room temperature.
  Interventions: Dietary Supplement: Tap water

INTERVENTIONS:
Dietary Supplement: "Acqua Santa di Chianciano"® (sulphate-bicarbonate-calcium water) — During the first 4 weeks the SW-D patients will be asked to drink every morning, before breakfast, within 30 minutes, 500 mL of "Acqua Santa di Chianciano"® at room temperature.
  Arms: sulphate-bicarbonate-calcium water and low-calorie diet (SW-D)
Dietary Supplement: Tap water — During the first 4 weeks the TW-D patients will be asked to drink every morning, before breakfast, within 30 minutes, 500 mL of tap water at room temperature.
  Arms: tap water and low-calorie diet (TW-D)

SUMMARY:
Overweight and obese patients will be recruited and randomly assigned to two groups of intervention. To the first group [sulphate-bicarbonate-calcium water and low-calorie diet (SW-D)] will be administered "Acqua Santa di Chianciano"®, associated to a personalized low calorie diet, while the second group [tap water and low-calorie diet (TW-D)] will follow the personalized low calorie diet but will be asked to drink the same quantity of tap water, over a 4 week period. Stool samples will be collected and analyzed for changes in gut microbiota composition. Patients' body weight will be recorded at the beginning and at the end of the study.

DETAILED DESCRIPTION:
Overweight (BMI>25) and obesity in adults is a global public health concern because weight excess increases the relative risk of disease and mortality 1-4. A range of diseases, notably cardiovascular disease, diabetes and a number of cancers, are related to excess weight 5. Traditional low-calorie diets are frequently ineffective 6. Although a number of pharmacological approaches for treatment of obesity have been investigated, only few are safe and most of them have adverse effects 7,8. Thus, further studies are necessary in order to find natural antiobesity remedies. Gut microbiota composition is thought to influence body weight 9.

As recently demonstrated in our previous study 10, "Acqua Santa di Chianciano"® helps to maintain the body weight and the values of serum lipids stable in subjects under a relatively high-calorie diet. Possible mechanisms may be a) changing the gut microbiota composition and/or b) increasing the concentration and/or the qualitative pattern of serum bile acids with a subsequent increase of the energy expenditure 11. This study wants to assess the effectiveness in losing weight of "Acqua Santa di Chianciano"® in addition to a low-calorie diet and its effects on gut microbiota composition.

ELIGIBILITY:
Inclusion Criteria:

* Women with BMI between 29 and 35 kg/m2
* Age between 18 and 65 years

Exclusion Criteria:

* Therapy with antibiotics, bile salts, cholestyramine, laxatives, pre- or probiotics during the last 3 months before enrollment
* Helycobacter Pylori positivity
* Previous cholecystectomy
* Gallbladder disease
* Cholestasis
* Consumption of more than 20 g of alcohol/day
* Inflammatory bowel diseases
* Previous gastrointestinal surgery modifying the anatomy
* Pregnancy or lactating state
* Prescribed hypocaloric diet in the three previous months

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2020-11-19 (Actual)

PRIMARY OUTCOMES:
weight loss | 12 weeks
  The primary end-point of the present study is to assess the effect on body weight of the association between sulphate-bicarbonate-calcium water consumption and low-calorie diet (SW-D) compared to tap water and the low-calorie diet (TW-D). The expected result is to obtain a 50% greater mean weight loss in the SW-D than in the TW-D group.

SECONDARY OUTCOMES:
gut microbiota composition | 4 weeks
  One of the secondary end-points is the evaluation of the effects of the association between low-calorie diet and sulphate-bicarbonate-calcium water consumption on gut microbiota.
body composition | 4 weeks
  One of the secondary end-points is the evaluation of the effects of the association between low-calorie diet and sulphate-bicarbonate-calcium water consumption on body composition (lean body mass/fat body mass) assessed by BIA.
bile acids pool | 4 weeks
  One of the secondary end-points is the evaluation of the effects of the association between low-calorie diet and sulphate-bicarbonate-calcium water consumption on the bile acids pool.
energy expenditure | 4 weeks
  One of the secondary end-points is the evaluation of the effects of the association between low-calorie diet and sulphate-bicarbonate-calcium water consumption on energy expenditure
thyroid function | 4 weeks
  One of the secondary end-points is the evaluation of the effects of the association between low-calorie diet and sulphate-bicarbonate-calcium water consumption on thyroid function

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Ginanni Corradini, MD, PhD, Study Director — Department of Clinical Medicine, Sapienza University of Rome, Umberto I Hospital; Fredrik Bäckhed, PhD, Study Director — Wallenberg Laboratory, SU/Sahlgrenska, SE-413 45 Göteborg, Sweden; Alessandro Laviano, MD, PhD, Principal Investigator — Department of Translational and Precision Medicine, Sapienza University of Rome; Lorenzo Maria Donini, MD, Principal Investigator — Department of Experimental Medicine, Sapienza University of Rome; Adriano De Santis, MD, Principal Investigator — Department of Translational and Precision Medicine, Sapienza University of Rome; Maurizio Muscaritoli, MD, Principal Investigator — Department of Translational and Precision Medicine, Sapienza University of Rome; Isabella Preziosa, MD, Principal Investigator — Department of Translational and Precision Medicine, Sapienza University of Rome
Locations (1):
- Department of Translational and Precision Medicine, Sapienza University of Rome, Rome, Italy

REFERENCES:
- [Background] Flegal KM, Graubard BI, Williamson DF, Gail MH. Excess deaths associated with underweight, overweight, and obesity. JAMA. 2005 Apr 20;293(15):1861-7. doi: 10.1001/jama.293.15.1861. PMID 15840860
- [Background] Gronniger JT. A semiparametric analysis of the relationship of body mass index to mortality. Am J Public Health. 2006 Jan;96(1):173-8. doi: 10.2105/AJPH.2004.045823. Epub 2005 Aug 30. PMID 16131644
- [Background] Peeters A, Barendregt JJ, Willekens F, Mackenbach JP, Al Mamun A, Bonneux L; NEDCOM, the Netherlands Epidemiology and Demography Compression of Morbidity Research Group. Obesity in adulthood and its consequences for life expectancy: a life-table analysis. Ann Intern Med. 2003 Jan 7;138(1):24-32. doi: 10.7326/0003-4819-138-1-200301070-00008. PMID 12513041
- [Background] Sjostrom L. Review of the key results from the Swedish Obese Subjects (SOS) trial - a prospective controlled intervention study of bariatric surgery. J Intern Med. 2013 Mar;273(3):219-34. doi: 10.1111/joim.12012. Epub 2013 Feb 8. PMID 23163728
- [Background] Jeffery RW, Kelly KM, Rothman AJ, Sherwood NE, Boutelle KN. The weight loss experience: a descriptive analysis. Ann Behav Med. 2004 Apr;27(2):100-6. doi: 10.1207/s15324796abm2702_4. PMID 15026294
- [Background] Ryan DH, Bray GA, Helmcke F, Sander G, Volaufova J, Greenway F, Subramaniam P, Glancy DL. Serial echocardiographic and clinical evaluation of valvular regurgitation before, during, and after treatment with fenfluramine or dexfenfluramine and mazindol or phentermine. Obes Res. 1999 Jul;7(4):313-22. doi: 10.1002/j.1550-8528.1999.tb00414.x. PMID 10440587
- [Background] Carter R, Mouralidarane A, Ray S, Soeda J, Oben J. Recent advancements in drug treatment of obesity. Clin Med (Lond). 2012 Oct;12(5):456-60. doi: 10.7861/clinmedicine.12-5-456. PMID 23101148
- [Background] Greiner T, Backhed F. Effects of the gut microbiota on obesity and glucose homeostasis. Trends Endocrinol Metab. 2011 Apr;22(4):117-23. doi: 10.1016/j.tem.2011.01.002. Epub 2011 Feb 23. PMID 21353592
- [Background] Corradini SG, Ferri F, Mordenti M, Iuliano L, Siciliano M, Burza MA, Sordi B, Caciotti B, Pacini M, Poli E, Santis AD, Roda A, Colliva C, Simoni P, Attili AF. Beneficial effect of sulphate-bicarbonate-calcium water on gallstone risk and weight control. World J Gastroenterol. 2012 Mar 7;18(9):930-7. doi: 10.3748/wjg.v18.i9.930. PMID 22408352
- [Background] Watanabe M, Houten SM, Mataki C, Christoffolete MA, Kim BW, Sato H, Messaddeq N, Harney JW, Ezaki O, Kodama T, Schoonjans K, Bianco AC, Auwerx J. Bile acids induce energy expenditure by promoting intracellular thyroid hormone activation. Nature. 2006 Jan 26;439(7075):484-9. doi: 10.1038/nature04330. Epub 2006 Jan 8. PMID 16400329